CLINICAL TRIAL: NCT00610870
Title: Effect of Atorvastatin Administration Before Primary Percutaneous Coronary Intervention in Patients With ST-segment Elevation Myocardial Infarction
Brief Title: Effect of Atorvastatin Administration Before Primary Percutaneous Coronary Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: HC Gwon, MD,PhD / Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-04-049
Record Dates: First submitted 2008-01-27; First posted 2008-02-08 (Estimated); Last update posted 2011-03-03 (Estimated); Status verified 2011-03

CONDITIONS: Angioplasty, Transluminal, Percutaneous Coronary
Keywords: Myocardial infarct size; Atorvastatin; SPECT; Hydroxymethylglutaryl-CoA Reductase Inhibitors
MeSH Terms: interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Atorvastatin group
  Interventions: Drug: atorvastatin
- 2 (No Intervention): Control group

INTERVENTIONS:
Drug: atorvastatin — atorvastatin 80mg/day before primary coronary intervention
  Arms: 1

SUMMARY:
The purpose of this study to determine whether statin pretreatment decrease myocardial infarct size in patients with acute myocardial infarction undergoing primary percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

* Presence of chest pain for more than 30 minutes but less than 12 hours after symptom onset
* ST segment elevation more than 1 mm in two or more contiguous leads or presumably a new onset left bundle branch blockage

Exclusion Criteria:

* Cardiogenic shock
* History of myocardial infarction
* Chronic liver disease
* Previous or current statin use

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2007-07; Primary Completion 2009-02 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Myocardial infarct size by SPECT | between 5 and 14 days after acute myocardial infarction

SECONDARY OUTCOMES:
Myocardial infarct size measured by contrast-enhanced MRI | within 14 days after acute myocardial infarction
Myocardial blush grade after the procedure | immediate after procedure
complete ST resolution | at 60 minutes after the procedure
major adverse cardiac events related to left ventricular dysfunction (death, new-onset sustained hypotension or heart failure, and hospital readmission for left ventricular dysfunction) | at 6 months after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Hyeon-Cheol Gwon, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea